CLINICAL TRIAL: NCT03085563
Title: A Comparison of Intranasal Midazolam and Nitrous Oxide (N2O) Minimal Sedation for Minor Procedures in a Pediatric Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-1909
Record Dates: First submitted 2016-10-21; First posted 2017-03-21 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Conscious Sedation; Simple Lacerations Less Than 4 cm; Lumbar Punctures; Minor Incision Drainage of Abscesses Not Requiring Extensive Debridement
MeSH Terms: interventions — Nitrous Oxide; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Oxide (Active Comparator): Nitrous oxide will be delivered in one of two ways, using the titration method or rapid infusion method.
  Interventions: Drug: Nitrous Oxide
- Intranasal Midazolam (Active Comparator): Intranasal midazolam with mucosal atomizer device administration will follow the Children's Hospital Colorado (CHCO) established policy 'Intranasal Administration (atomization) of Medications'.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous oxide will be delivered in one of two ways, using the titration method or rapid infusion method. Which ever method is used will be recorded. When using the titration method, starting at 20%, nitrous oxide will be added in 10% increments every 60 seconds until the ideal level of sedation has been met (not to exceed 70% nitrous oxide). Using the rapid infusion method, after the proper flow rate has been achieved with oxygen, the flowmeter will be increased to obtain 50% concentration of nitrous oxide. After 2-3 minutes if the patient does not have adequate sedation, nitrous oxide concentration will be increased to 70%.
  Other Names: N2O
  Arms: Nitrous Oxide
Drug: Midazolam — Intranasal midazolam with mucosal atomizer device administration will follow the Children's Hospital Colorado (CHCO) established policy 'Intranasal Administration (atomization) of Medications'. As per standard of care, each patient will receive a standardized dose of 0.4mg/kg (maximum dose of 10mg) of intranasal midazolam with the mucosal atomizer device for all procedures.
  Other Names: Versed
  Arms: Intranasal Midazolam

SUMMARY:
The objective of this project is to compare the sedative effects of intranasal midazolam versus inhaled nitrous oxide (N2O) for minor procedures in the pediatric emergency department. The primary outcome will be length of stay (LOS) in the emergency department (ED) stay for minor procedures. Secondarily the investigators will compare patient/family and provider satisfaction while using either intranasal midazolam or N2O for minimal sedation. The investigators hypothesize that the total length of stay for children undergoing minor procedures in the ED will be lower for N2O, as compared to intranasal midazolam. The investigators also hypothesize that patient/family and provider satisfaction will be higher with N2O and adverse effects will not differ between N2O and intranasal midazolam. Patients will receive either intranasal midazolam or N2O for minor procedures. Following the enrollment period, data will be analyzed and the two will be compared. Total length of stay, patient/family and provider satisfaction will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥2 years of age and <18 years of age, and
2. Parent/legal guardian age ≥18 years of age to <80 years of age
3. Patients with an American Society of Anesthesiologists (ASA) Physical Status Classification System level 1, 2, and 3
4. Patients requiring anxiolysis and mild sedation for minor procedures

   1. Minor procedures will include simple lacerations less than 4 cm
   2. Lumbar punctures
   3. Minor incision
   4. Drainage of abscesses that do not require extensive debridement
5. Must receive the standard of care dosing for either nitrous oxide or intranasal midazolam.

   1. Nitrous oxide up to 70% nitrous concentration will be allowed
   2. Intranasal Midazolam 0.4mg/kg with a max dose of 10mg

Exclusion Criteria:

1. Nasal injury, nasal obstruction or significant congestion
2. Laceration that involves the nose and ears or come into contact with the scavenger device or nitrous oxide tubing
3. Allergy to benzodiazepines
4. Benzodiazepine dosing for any reason 24 hours prior to procedure
5. Excessive Epistaxis
6. Facial or nasal deformity
7. Copious mucous
8. Recent (less than 1 week) tympanic membrane graft or middle ear surgery
9. Recent bleomycin therapy
10. Patients known to be pregnant at time of enrollment
11. Patients with severe behavior problems, personality disorders or other mind-altering conditions as determined by administering provider.
12. Closed space situations such as:

    1. pneumothorax,
    2. air embolus,
    3. pneumocephalus, or
    4. craniotomy in the last 3 weeks,
    5. intraocular surgery with retained gas,
    6. pulmonary bullae,
    7. severe emphysema, or
    8. bowel obstruction.
13. Patients with significant co-morbidities:

    1. severe pulmonary disease,
    2. cardiac disease,
    3. hematologic diseases associated with B12 deficiency,
    4. sickle cell disease.
14. Patients with acute otitis media and/or sinusitis
15. History of paradoxical reaction to nitrous oxide
16. Known Methicillin-resistant Staphylococcus aureus (MRSA+) patients
17. Co-administration of additional sedation or analgesic medications

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Szefler, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were excluded prior to randomization (two withdrawals, one screen failure).
Period: Overall Study
Arm/Group | Nitrous Oxide | Intranasal Midazolam
Started | 19 | 41
Completed | 19 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrous Oxide | Intranasal Midazolam | Total
Number analyzed (Participants) | 19 | 41 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 41 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 7 | 28 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 41 | 60

OUTCOME MEASURES:

1. Primary Outcome: ED Length of Stay After Intranasal Midazolam or Nitrous Oxide Administration
Description: The total length of Emergency Department (ED) stay will be defined as time from intranasal midazolam or nitrous oxide administration to time of discharge readiness, collected by the research assistants. Additional time periods measured will include: time from anxiolytic/sedative given to time of procedure completion, and total time for recovery.
Time Frame: From administration of intranasal midazolam or nitrous oxide, assessed over an estimated time of 2 hours.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Nitrous Oxide | Intranasal Midazolam
Number analyzed (Participants) | 19 | 41
minutes
  Time from intranasal midazolam or nitrous oxide administration to time of discharge readiness | 24.5 [15.5 to 33.5] | 18.5 [16 to 34]
  Time from anxiolytic/sedative given to time of procedure completion | 9 [3 to 19] | 10 [6 to 16]
  Total time for recovery | 15.5 [12.5 to 17.5] | 8.5 [7 to 18]

2. Secondary Outcome: Patient/Parent and Provider Satisfaction With Sedation and Anxiolytic/Sedative.
Description: Patient/parent satisfaction will be assessed for all patients; child satisfaction will be assessed for patients over 12 years of age. Satisfaction will be measured on a scale of 1 to 5 (1 being not satisfied and 5 being very satisfied). Specifically, parents (and children when applicable) will be asked "how satisfied with the means of sedation were you for the procedure performed". Research assistants will then ask the ED providers on a scale of 1 to 5 (1 being not satisfied and 5 being very satisfied) "how satisfied with the means of sedation were you for the procedure performed".
Time Frame: Time of discharge, Approximately 2 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Nitrous Oxide | Intranasal Midazolam
Number analyzed (Participants) | 19 | 41
score on a scale
  Parent/Patient | 5 [5 to 5] | 5 [4 to 5]
  Provider | 5 [4 to 5] | 4.5 [4 to 5]

3. Secondary Outcome: Adverse Events.
Description: Number of adverse events observed. Adverse events will be classified and defined as hypoxia, need for administration of reversal agent, nausea, vomiting, paradoxical reaction, airway obstruction, laryngospasm, inadequate sedation, allergic reaction, and cardiac arrest.
Time Frame: Time of discharge, Approximately 2 hours
Measure: Number; unit: Adverse Events
Arm/Group | Nitrous Oxide | Intranasal Midazolam
Number analyzed (Participants) | 19 | 41
Adverse Events
  hypoxia | 0 | 3
  need for administration of reversal agent | 0 | 0
  nausea, vomiting | 0 | 0
  paradoxical reaction | 0 | 1
  airway obstruction | 0 | 0
  laryngospasm | 0 | 0
  inadequate sedation | 0 | 0
  allergic reaction | 0 | 0
  cardiac arrest | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Nitrous Oxide | Intranasal Midazolam
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/41
Other Adverse Events (participants affected / at risk) | 0/19 | 4/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrous Oxide (N=19) | Intranasal Midazolam (N=41)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
paradoxical reaction (Nervous system disorders) | 0 (0) | 1 (1) — Product made participant more agitated/anxious

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03085563/Prot_SAP_000.pdf